CLINICAL TRIAL: NCT02663791
Title: Alcohol Consumption and Arterial Stiffness: A Longitudinal Study of Pulse Wave Velocity in the Whitehall II Cohort
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); Alcohol Research UK (Other)
Responsible Party: Principal Investigator, Dara O'Neill, Research Associate, University College, London
Other Study IDs: Whitehall II - Alcohol PWV 01
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aortic Stiffness
Keywords: Alcohol; Aortic stiffness; Arterial stiffness; Pulse wave velocity; Longitudinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Arterial stiffness is an important marker of cardiovascular health. Recent evidence from cross-sectional research has suggested it is associated with alcohol consumption. Research that employs a longitudinal perspective may be better equipped to evaluate the nature of this relationship and in particular to determine whether alcohol consumption is linked to the progression of arterial stiffness over time. The current study will consequently implement a longitudinal cohort design to evaluate the association between long-term alcohol consumption patterns and changes in arterial stiffness. Data will be drawn from the Whitehall II cohort study of British civil servants, in which participants completed repeat pulse wave velocity (PWV) assessments of arterial stiffness across a four-to-five year interval. Repeat measurements of volume of alcohol intake were also recorded for participants, extending back across more than two decades. Intake will be categorised in such a way as to distinguish between different alcohol consumer types, including non-drinkers and former drinkers. Linear mixed effects models will be used with adjustment for potential confounds, such as age, diabetes, mean arterial pressure and heart rate. Results from the modelling work will illustrate the extent and form of the association between alcohol intake and PWV. This work will provide useful insights into the role that alcohol intake plays in the longitudinal progression of an important cardiac marker, and it will have implications for our understanding of alcohol's relationship to cardiovascular health in the general population.

DETAILED DESCRIPTION:
Arterial stiffness occurs where the vessel wall lacks elasticity. It is known to be independently associated with both cardiovascular morbidity and mortality, such that it can act as a surrogate end point for studies of cardiovascular disease. Pulse wave velocity (PWV) is an index of this stiffness and has been described as its 'gold standard' measurement.

A number of other clinical factors have been found to show meaningful association with PWV, including heart rate and mean arterial pressure. These findings have highlighted the need for studies of new potential determinants of PWV to account for the potentially confounding influence of these known factors. Additional demographic and lifestyle characteristics have also been shown to act as moderators of PWV. In particular, research has demonstrated that PWV increases with age, and this stiffness is consequently deemed an indicator of vascular ageing.

Alcohol intake is another lifestyle characteristic that has been considered as a potential factor in the loss of arterial elasticity. Evidence to date suggests that a J-shaped association may exist between such intake and PWV, but this work has mostly relied on cross-sectional data or looked at short-term intake patterns only. By adopting a longitudinal perspective, further insight may be garnered into this important epidemiological issue. Consequently, the new study herein proposed will address this research need and investigate how different patterns of alcohol consumption relate to arterial stiffness and to the progression of this stiffness over time. The primary objectives of this study are to (1) examine whether long-term patterns of alcohol consumption are independently associated with a baseline assessment of carotid-femoral PWV and (2) whether alcohol intake is likewise associated with longitudinal changes in this important cardiovascular marker.

Longitudinal alcohol exposure will be determined from reported consumption at phases 1 (1985-1988) through 9 (2007-2009) of the Whitehall II Cohort Study and categorised according to the latest UK recommendations on alcohol intake limits. These guidelines define moderate consumption as weekly ethanol intake volumes of 112g or under for both males and females. As alcohol consumption is recorded in UK units in the Whitehall II database, conversion will be performed using the standard ratio of 1 unit to 8 grams of ethanol prior to categorisation. The subsequent categorisation will draw distinctions between non-drinkers and former drinkers, as well as between moderate and heavy consumers. Those with unstable patterns of consumption will also be identified as there is emerging evidence that such consumers may have a different cardiovascular risk profile compared to consumers with more longitudinally consistent intake patterns.

Demographic and clinical characteristics will be investigated to provide context for the subsequent inferential analyses. As research has also suggested that participant sex can moderate the relationship between alcohol and PWV, this will be tested in the current analysis (through preliminary modelling that includes sex as part of an interaction term with level of alcohol consumption). If this moderation effect is replicated, then our core result reporting will be stratified according to sex.

Linear mixed effects models will then be used to examine the effect of long-term alcohol consumption on PWV and its effect on subsequent longitudinal changes in this cardiovascular marker. This modelling approach is particularly suited to analysing the complex data structure under investigation, including the correlation across individual participants' paired measurements. A detailed analytic protocol is available upon request.

Supplementary linear mixed effects modelling will also be performed to look at the association between short-term alcohol consumption patterns and PWV. This will employ the same modelling strategy as used in the primary analysis above, with the categorisation of consumption utilising reported intake at the most recent assessment phase only. This supplementary analysis will offer additional context for the findings of the primary analysis and provide further detail on the relationship that different forms of alcohol consumption have with arterial stiffness.

Through this comprehensive and detailed analysis, it is hoped that new insights on this important issue of cardiovascular health will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Whitehall II cohort study
* Reported alcohol consumption on a minimum of one occasion between phase 1 and phase 9 of the Whitehall II cohort study

Exclusion Criteria:

* Left Whitehall II cohort study prior to phase 9 or did not participate in PWV assessment at Phase 9
* Had history of coronary heart disease

Ages: 34 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be drawn from the Whitehall II cohort study database. This incorporates longitudinal assessments of 6,895 male (67%) and 3,413 female British civil servants, originally recruited between 1985 and 1988. The overall age range was 34 to 56 years. Of these, 897 were excluded due to having a history of cardiovascular disease. Clinical assessments were repeated at 4-to-5 year intervals. PWV measurement was introduced to the protocol at phase 9, with assessments taking place during 2008 and 2009. 3,869 of the sample participants had a successful PWV assessment during this time. Follow-up testing took place at phase 11, during 2012 and 2013. Of the participants who underwent a PWV assessment at phase 9, 3,130 also had a successful PWV assessment at phase 11. This group included 2,350 males (75%) and 780 females.
Sampling Method: Non-Probability Sample
Enrollment: 10308 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Baseline Carotid-Femoral Pulse Wave Velocity | 1 day
  A baseline carotid-femoral pulse wave velocity (PWV) assessment occurred at phase 9 (each participant attended an assessment day during 2008 or 2009) of the Whitehall II cohort study. Up to 3 PWV measurements were performed during this assessment, and where a participant underwent multiple measurements, the mean of these will be calculated for that participant and used as their baseline PWV measurement.
Change from Baseline Carotid-Femoral Pulse Wave Velocity at Follow-Up | 4 to 5 years
  Change in carotid-femoral PWV between the baseline and follow-up PWV assessments will be investigated. The follow-up PWV assessment occurred at phase 11 (2012-2013) of the Whitehall II cohort study. Up to 3 PWV measurements were again performed during this assessment, and where a participant underwent multiple measurements, the mean of these will be calculated for that participant and used as their follow-up PWV measurement.

CONTACTS AND LOCATIONS:
Overall Officials: D O'Neill, PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can request access to anonymised data: http://www.ucl.ac.uk/whitehallII/data-sharing

REFERENCES:
- [Background] Marmot M, Brunner E. Cohort Profile: the Whitehall II study. Int J Epidemiol. 2005 Apr;34(2):251-6. doi: 10.1093/ije/dyh372. Epub 2004 Dec 2. No abstract available. PMID 15576467
- [Background] Cavalcante JL, Lima JA, Redheuil A, Al-Mallah MH. Aortic stiffness: current understanding and future directions. J Am Coll Cardiol. 2011 Apr 5;57(14):1511-22. doi: 10.1016/j.jacc.2010.12.017. PMID 21453829
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Cecelja M, Chowienczyk P. Role of arterial stiffness in cardiovascular disease. JRSM Cardiovasc Dis. 2012 Jul 31;1(4):cvd.2012.012016. doi: 10.1258/cvd.2012.012016. PMID 24175067
- [Background] Cecelja M, Chowienczyk P. Dissociation of aortic pulse wave velocity with risk factors for cardiovascular disease other than hypertension: a systematic review. Hypertension. 2009 Dec;54(6):1328-36. doi: 10.1161/HYPERTENSIONAHA.109.137653. Epub 2009 Nov 2. PMID 19884567
- [Background] Matsumoto C, Tomiyama H, Yamada J, Yoshida M, Shiina K, Nagata M, Yamashina A. Association of blood pressure levels with the effects of alcohol intake on the vasculature in Japanese men. Hypertens Res. 2009 Feb;32(2):127-32. doi: 10.1038/hr.2008.23. Epub 2009 Jan 16. PMID 19262471
- [Background] Beilin L. Alcohol and cardiovascular disease: possible protection via effects on aortic stiffness. J Hypertens. 2005 Apr;23(4):703-5. doi: 10.1097/01.hjh.0000163133.62020.98. No abstract available. PMID 15775769
- [Background] Sasaki S, Yoshioka E, Saijo Y, Kita T, Okada E, Tamakoshi A, Kishi R. Relation between alcohol consumption and arterial stiffness: A cross-sectional study of middle-aged Japanese women and men. Alcohol. 2013 Dec;47(8):643-9. doi: 10.1016/j.alcohol.2013.10.003. Epub 2013 Oct 17. PMID 24239150
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Derived] O'Neill D, Britton A, Brunner EJ, Bell S. Twenty-Five-Year Alcohol Consumption Trajectories and Their Association With Arterial Aging: A Prospective Cohort Study. J Am Heart Assoc. 2017 Feb 20;6(2):e005288. doi: 10.1161/JAHA.116.005288. PMID 28219925
- See also: UCL Research Department of Epidemiology & Public Health — https://www.ucl.ac.uk/epidemiology